CLINICAL TRIAL: NCT00752674
Title: The Effectiveness of Neuromuscular Balance in Low Back Pain
Brief Title: Neuromuscular Balance in Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fortaleza University (Other)
Responsible Party: Karla Adryana Diniz Meireles, Fortaleza University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 265-2006
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2008-09-15 (Estimated); Status verified 2008-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; physical therapy; pain
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Neuromuscular balance
  Interventions: Other: Neuromuscular balance

INTERVENTIONS:
Other: Neuromuscular balance

SUMMARY:
The research was an interventional study with a quantitative board, fulfilled in a private clinique specialized in trauma service; it was formed between august to October of 2006. The objective was to investigate the effectiveness of neuromuscular balance in lumbar pain. The 12 patients, with age between 20 and 55 years, whose did five consultations, with 100% presence, got relief of the pain and increase of movement of hips' articulation which was the most painful movement with 91,66% graduation. All the patients presented the shorting test positive and it kept positive in 7 patients. There was a significant improvement in pain relief (p=0,001,) comparing the first and the fifth consultation, and hip articulation movement. Even after the relief of the pain, 7(58,3%) of the patients kept the treatment for a more effective rehabilitation and prevention of repetition of the symptoms. It was concluded that the neuromuscular balance relieved quickly the pain, being essential for effective rehabilitation of low back pain, with the inclusion of others manual techniques.

DETAILED DESCRIPTION:
The low back pain is a symptom presented in muscle-skeletal change on lumbar region, preferring young adults, in economic active fase. The neuromuscular balance was developed by Soulier when he met the "activator methods" which was a pen that create vibrations and consist in a vibration or a micro thrust to reduce the articulation and spinal problems through a non manipulative correction. The research was un interventional study with a quantitative board, fulfilled in a private clinique specialized in trauma service; it was formed between august to October of 2006. The objective was to investigate the effectiveness of neuromuscular balance in lumbar pain. The 12 patients, with age between 20 and 55 years, whose did five consultations, with 100% presence, got relief of the pain and increase of movement of hips' articulation which was the most painful movement with 91,66% graduation. All the patients presented the shorting test positive and it kept positive in 7 patients. There was a significant improvement in pain relief (p=0,001,) comparing the first and the fifth consultation, and hip articulation movement. Even after the relief of the pain, 7(58,3%) of the patients kept the treatment for a more effective rehabilitation and prevention of repetition of the symptoms. It was concluded that the neuromuscular balance relieved quickly the pain, being essential for effective rehabilitation of low back pain, with the inclusion of others manual techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low back pain between 20 and 55 years old, submitted to a physical therapy treatment.

Exclusion Criteria:

* Patients with no miofascial low back pain

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2006-08; Primary Completion 2006-10 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karla Adryana Diniz Meireles, Master, Principal Investigator — Fortaleza University